CLINICAL TRIAL: NCT05163041
Title: Phase 1/2 Study of the Safety, Pharmacokinetics, and Preliminary Clinical Activity of BT7480 in Patients With Nectin-4 Associated Advanced Malignancies
Brief Title: Study BT7480-100 in Patients With Advanced Malignancies Associated With Nectin-4 Expression
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BicycleTx Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT7480-100
Record Dates: First submitted 2021-11-19; First posted 2021-12-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BT7480 monotherapy dose escalation (Experimental): Participants will receive increasing doses of BT7480. It is expected that approximately 80 patients will participate in this dose escalation arm.
  Interventions: Drug: BT7480
- BT7480 and nivolumab dose escalation (Experimental): Participants will receive increasing doses of BT7480 and standard dose of nivolumab. It is expected that approximately 12 patients will participate in this dose escalation arm.
  Interventions: Drug: BT7480; Drug: Nivolumab
- BT7480 monotherapy dose expansion (Experimental): Participants will receive a selected dose of BT7480. It is expected that approximately 45 patients will participate in this dose expansion arm in Phase 2.
  Interventions: Drug: BT7480
- BT7480 and nivolumab dose expansion (Experimental): Participants will receive a selected dose of BT7480 and standard dose of nivolumab. It is expected that approximately 45 patients will participate in this dose expansion arm in Phase 2.
  Interventions: Drug: BT7480; Drug: Nivolumab
- BT7480 monotherapy in patients with renal insufficiency (Experimental): Participants will receive a selected dose of BT7480. It is expected that approximately 12 patients will participate in this dose confirmation arm.
  Interventions: Drug: BT7480

INTERVENTIONS:
Drug: BT7480 — Participants will receive a 60 minute IV infusion of BT7480 once weekly (i.e., on Days 1,8,15 and 22) during a 28-day cycle
Drug: Nivolumab — Nivolumab will be given as a 240mg dose every 2 weeks administered as per local labelling as a 30 minute IV infusion
  Arms: BT7480 and nivolumab dose escalation; BT7480 and nivolumab dose expansion

SUMMARY:
This clinical study is evaluating a drug called BT7480 alone and in combination with nivolumab in participants with advanced solid tumors associated with Nectin-4 expression.

The main goals of the study are to:

* Find the recommended dose of BT7480 that can be given safely to participants alone and in combination with nivolumab
* Learn about the side effects and effectiveness of BT7480 alone and in combination with nivolumab
* Learn about the effect BT7480 has on the body and how BT7480 is cleared by the body
* Learn about the side effects and effectiveness of BT7480 in patients with reduced kidney function

DETAILED DESCRIPTION:
BT7480 is a tumor targeted immune cell agonist consisting of three bicyclic peptides (Bicycle®) conjugated via a linker, one that binds selectively to Nectin-4 and two that bind to CD137.

This study is a Phase 1/2, multicenter, first-in-human, open-label study of BT7480 given as a single agent and in combination with nivolumab once weekly. There are five parts to the trial: 1) Phase 1 dose escalation in patients with select advanced solid tumors primarily to evaluate safety and tolerability of BT7480 as a monotherapy and determine a recommended Phase 2 dose (RP2D); 2) Phase 1 dose escalation in combination with nivolumab, once the monotherapy RP2D has been determined; 3) Phase 2 dose expansion as a monotherapy once the RP2D has been determined; 4) Phase 2 dose expansion in combination with nivolumab; 5) Phase 1 monotherapy dose confirmation in patients with renal insufficiency once the monotherapy RP2D has been determined

ELIGIBILITY:
Inclusion Criteria:

* Must have locally advanced or metastatic disease that is refractory to standard therapy, or for which no standard therapy is judged to be appropriate or provide clinical benefit, as judged by the Investigator
* Must have a histologically or cytologically confirmed malignant solid tumor associated with Nectin-4 expression, including, but not limited to, urothelial (transitional cell) carcinoma; head and neck squamous cell carcinoma; non-small cell lung cancer; and ovarian, breast, gastric, or esophageal carcinoma
* Must have ECOG performance status score 0 or 1 and acceptable organ and hematological function
* Must have metastatic or locally advanced disease and measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Life expectancy ≥12 weeks
* Must submit fresh or archival tumor tissue
* Must provide written informed consent, according to local guidelines, signed and dated by the patient or by a legal guardian prior to the performance of any study-specific procedures, sampling, or analysis

Exclusion Criteria:

* Prior therapy with a cytotoxic, small molecule, or other systemic chemotherapy within 14 days of the first dose of study drug
* Prior immunotherapy, including monoclonal antibodies, within 28 days or 5 half-lives of the first dose of study drug, whichever is shorter
* Prior treatment with CD137 targeted therapy
* Mean resting QTc (eg, QTcF) greater than 470 msec on triplicate electrocardiograms (ECGs) obtained at screening
* Uncontrolled symptomatic brain metastases
* Uncontrolled diabetes with glycosylated hemoglobin greater than or equal to 8%
* Uncontrolled hypertension at screening or prior to initiation of study drug
* History of autoimmune disease except well-controlled diabetes mellitus, alopecia, well controlled thyroid disease or vitiligo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment emergent adverse events in dose escalation phase | From Cycle 1 Day 1 (each cycle is 28 days) until 30 (+/-5) days after the last dose of study drug
  Incidence and severity of treatment emergent adverse events to assess safety and tolerability following treatment with BT7480 alone and in patients with renal insufficiency using NCI CTCAE v5.0 criteria
Number of patients with treatment emergent adverse events in dose escalation phase | From Cycle 1 Day 1 (each cycle is 28 days) until 125 (+/-5) days after the last dose of study drug
  Incidence and severity of treatment emergent adverse events to assess safety and tolerability following treatment with BT7480 and in combination with nivolumab using NCI CTCAE v5.0 criteria
Confirmed response rate as measured by overall response rate (ORR) to demonstrate clinical activity following treatment with BT7480 in dose expansion phase | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Overall response rate (ORR) following treatment with BT7480 alone and in combination with nivolumab according to RECIST 1.1 criteria nivolumab according to RECIST 1.1 criteria
Confirmed response rate as measured by clinical benefit rate (CBR) to demonstrate clinical activity following treatment with BT7480 in dose expansion phase | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Clinical benefit rate (CBR) following treatment with BT7480 alone and in combination with nivolumab according to RECIST 1.1 criteria nivolumab according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Confirmed response rate as measured by overall response rate (ORR) to demonstrate clinical activity following treatment with BT7480 in dose escalation phase | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Overall response rate (ORR) following treatment with BT7480 alone and in combination with nivolumab and in patients with renal insufficiency according to RECIST 1.1 criteria
Confirmed response rate as measured by clinical benefit rate (CBR) to demonstrate clinical activity following treatment with BT7480 in dose escalation phase | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Clinical benefit rate (CBR) following treatment with BT7480 alone and in combination with nivolumab and in patients with renal insufficiency according to RECIST 1.1 criteria
Number of patients with treatment emergent adverse events in dose expansion phase | From Cycle 1 Day 1 (each cycle is 28 days) until 30 (+/-5) days after the last dose of study drug
  Incidence and severity of treatment emergent adverse events to assess safety and tolerability following treatment with BT7480 alone using NCI CTCAE v5.0 criteria
Number of patients with treatment emergent adverse events in dose expansion phase | From Cycle 1 Day 1 (each cycle is 28 days) until 125 (+/-5) days after the last dose of study drug
  Incidence and severity of treatment emergent adverse events to assess safety and tolerability following treatment with BT7480 alone using NCI CTCAE v5.0 criteria
Duration of response to assess clinical activity in dose escalation and dose expansion phase | From initial response to therapy to subsequent disease progression, an average of 6 months
  Duration of response following treatment with BT7480 alone and in combination with nivolumab and in patients with renal insufficiency
Progression free survival time in dose escalation and dose expansion phase | At 6 months
  Duration of time from first drug administration to disease progression according to RECIST 1.1 following treatment with BT7480 alone and in combination with nivolumab and in patients with renal insufficiency
Maximum plasma concentration (Cmax) of BT7480 | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Maximum plasma concentration (Cmax) of BT7480 in all participants receiving BT7480 alone or in combination with nivolumab
Area under the plasma concentration-time curve (AUC) of BT7480 | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Area under the plasma concentration-time curve (AUC) of BT7480 in all participants receiving BT7480 alone or in combination with nivolumab
Terminal half life (t1/2) of BT7480 in plasma | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Terminal half life (t1/2) of BT7480 in plasma in all participants receiving BT7480 alone or in combination with nivolumab
Cumulative amount of BT7480 excreted in the urine | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Cumulative amount of BT7480 excreted in the urine in all participants receiving BT7480 alone or in combination with nivolumab
Number of participants positive for anti-drug antibodies (ADA) | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Incidence of ADAs in patients treated with BT7480 alone or in combination with nivolumab
Level of CD137 target engagement in all patients | From Cycle 1 Day 1 (each cycle is 28 days) through study completion, an average of 6 months
  Level of CD137 target engagement in peripheral blood in patients treated with BT7480 alone or in combination with nivolumab

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - State University of Iowa, Iowa City, Iowa
  - Columbia University Irving Medical Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - START Center for Cancer Care, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: No